CLINICAL TRIAL: NCT04346875
Title: Is the Number of Dressing Changes Associated With Acute PJI Following Total Joint Arthroplasty? A Randomized Clinical Trial
Brief Title: Changing of Dressing for Periprosthetic Joint Infection in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, Residents Doctor in Orthopedics Department, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 30042020.02
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Infection; Surgical Site Infection; Prosthetic Infection; Wound Infection
MeSH Terms: conditions — Infections; Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Intervention Model Description: Single-blind
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regularly changing group (Experimental): Participants will undergo dressing every 3 days by the senior wound care nurse
  Interventions: Procedure: Regularly changing of dressing
- Non-changing group (Active Comparator): Participants will not be subject to dressing change.
  Interventions: Procedure: No application

INTERVENTIONS:
Procedure: Regularly changing of dressing — Conventional dressing
  Arms: Regularly changing group
Procedure: No application — No dressing change
  Arms: Non-changing group

SUMMARY:
The primary aim of the study is to compare two methods for a relationship with total knee infection: regular changing of dressings and not changing dressings.

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) is one of the most dreaded complications that occur after total joint arthroplasty. Periprosthetic joint infection remains an uncommon yet devastating complication that continues to influence the outcome of total joint arthroplasty. (1-4) Although different dressing methods have been described, the effect of changing the frequency of conventional dressings on PJI is curious.

After obtaining informed consent from all participants, parallel-group randomization will be performed with the help of a computer. The first dressing of all participants will be done in the operating room using the same materials. No drains will be used in any patient.

Then, according to the randomization, the procedures will be adjusted by the wound care nurse with the patient. All on-study and outcome data will be collected by the study staff blinded to study group assignment. The dressing group participants will be dressed by the same wound care nurse during the discharge. The dressing group participants will be dressed by the same wound care nurse in an outpatient service every three days using the same material. The total dressing number will be in the dressing group participant 5 times. Both group participants will be evaluated in the outpatient service after 2 weeks. Subsequently, all participants will be invited to check-in at the end of each month. All participants will be evaluated according to MSIS criteria in terms of superficial and deep periprosthetic infection.

The primary endpoint is to detect the difference between the incidence of periprosthetic infection after the regular dressing change and the incidence of the dressing unchanged group. In the secondary endpoint, it is to determine whether dressing change is an independent factor with multiple logistic regression test.

ELIGIBILITY:
Inclusion Criteria:

* Participants who agreed to inclusion in the study

Exclusion Criteria:

* Missing follow-up
* Participants with insufficient data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Periprosthetic infection rate | 90 days
  Incidence of patients to be diagnosed with periprosthetic infection according to MSIS criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Orkhan Aliyev, MD, Principal Investigator — Bezmialem Vakif University

IPD SHARING:
Plan to Share IPD: Yes
All IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Leta TH, Lygre SHL, Schrama JC, Hallan G, Gjertsen JE, Dale H, Furnes O. Outcome of Revision Surgery for Infection After Total Knee Arthroplasty: Results of 3 Surgical Strategies. JBJS Rev. 2019 Jun;7(6):e4. doi: 10.2106/JBJS.RVW.18.00084. PMID 31188156
- [Background] Berry DJ, Harmsen WS, Cabanela ME, Morrey BF. Twenty-five-year survivorship of two thousand consecutive primary Charnley total hip replacements: factors affecting survivorship of acetabular and femoral components. J Bone Joint Surg Am. 2002 Feb;84(2):171-7. doi: 10.2106/00004623-200202000-00002. PMID 11861721
- [Background] Soderman P, Malchau H, Herberts P. Outcome after total hip arthroplasty: Part I. General health evaluation in relation to definition of failure in the Swedish National Total Hip Arthoplasty register. Acta Orthop Scand. 2000 Aug;71(4):354-9. doi: 10.1080/000164700317393330. PMID 11028882